CLINICAL TRIAL: NCT01231139
Title: A Multi-centre Phase 2b Randomised Controlled Trial Investigating the Efficacy and Safety of Intravenous Paracetamol in Reducing Core Body Temperature After Traumatic Brain Injury
Brief Title: The Paracetamol AfteR Traumatic Brain InjurY Study
Acronym: PARITY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. M.K. Saxena (Other)
Collaborators: The George Institute (Other); The University of New South Wales (Other); Royal Brisbane and Women's Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Dr. M.K. Saxena, Intensive Care Physician, South East Sydney and Illawarra Area Health Service
Organization: South East Sydney and Illawarra Area Health Service (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PARITY
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Traumatic Brain Injury
Keywords: Brain Injury; Temperature; Paracetamol; Phase 2; TBI
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries | interventions — Acetaminophen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paracetamol (Experimental): Paracetamol dissolved in 0.9% Sodium Chloride
  Interventions: Drug: Paracetamol
- 0.9% Sodium Chloride (Placebo Comparator): 0.9% Sodium Chloride
  Interventions: Drug: 0.9% Sodium Chloride Schedule:

INTERVENTIONS:
Drug: Paracetamol — Intravenous paracetamol, 1 gram (100mls), administered over 30 minutes (every 4 hours for 3 days).
  Other Names: Perfalgan
  Arms: Paracetamol
Drug: 0.9% Sodium Chloride Schedule: — Identical placebo: 100mls saline given intravenous over 30 minutes (every 4 hours for 3 days)
  Other Names: Saline
  Arms: 0.9% Sodium Chloride

SUMMARY:
This primary aim is to investigate the effect of paracetamol in reducing body temperature in patients who have sustained traumatic brain injury. This study is also investigating the safety of paracetamol in this patient population.

DETAILED DESCRIPTION:
Traumatic head injury is a bruising of areas of the brain that occurs commonly as a result of a fall or a motor vehicle accident. Unfortunately, this is a common global occurrence and it occurs both in developing and developed countries. It causes death in nearly 1 in 3 of those who are most severely affected and a large proportion of those that survive have long-term physical or mental disability. Hence, traumatic head injury is a major global problem.

At present there are very few therapies that are known to be effective after a traumatic head injury. In particular the investigators are uncertain about whether modifying body temperature has any effect (good or bad) on the outcomes of patients. Although, this is practiced by some intensive care units around the world.

The investigators have searched extensively to look for any evidence that altering body temperature after traumatic head injury improves the outcome of patients (by reducing the amount of death or disability) and were unable to find any evidence at all. Some preliminary research in both animal experiments and clinical studies suggest that a raised temperature after forms of brain injury may in fact be harmful.

Therefore, at present the investigators believe that we do not really know what effect changing body temperature after head injury has on the outcome of patients.

The investigators are proposing to conduct a clinical study of patients who have had a severe head injury. The patients will be randomly allocated to 2 groups who will get either regular Paracetamol (dissolved in fluid) or a bottle of fluid without any Paracetamol. The 2 treatments will look identical and neither the patients nor the health care workers will know what treatment they are getting. Doing the study in this way will allow us to work out whether giving Paracetamol reduces the temperature of the body and whether there are any side effects that occur. If the study shows that Paracetamol can reduce body temperature safely in this setting then the investigators will work towards doing a larger study of treatments that reduce body temperature. The purpose of this larger study would be to see if the investigators can, not only reduce body temperature but also reduce amount of disability (physical and mental) as well as the death rate in traumatically brain injured patients.

In the proposed study the investigators will be using a higher dose of Paracetamol that is usually prescribed. Other research has shown that the dose that the investigators are proposing to use is safe and also that smaller doses in fact do not reduce body temperature.

ELIGIBILITY:
* Written informed consent has been obtained from the patient's next of kin
* Age > 18 and < 65
* Non penetrating head injury requiring mechanical ventilation, and, with an abnormal CT head (defined by the presence of haemorrhage, contusion, swelling, compression of basal cisterns or herniation)
* Within 72 hours of injury
* Presence (or imminent placement) of arterial cannula
* Alanine transferase level < 100

Exclusion Criteria:

* Suspected paracetamol overdose or allergy to paracetamol
* Confirmed or suspected pregnancy
* Use of pharmacological or physical intervention that reduces body temperature in the 6-hour period prior to randomisation.
* Clinician decision to institute any pharmacological or physical intervention that modifies body temperature
* Body temperature at time of recruitment less that 36°C or greater than 38.9°C
* History of chronic liver disease or chronic alcohol abuse
* Suspected malnutrition: BMI < 18 kg/m2 or weight < 60 kg
* BMI > 35 kg/m2
* Renal failure with serum creatinine > 200
* Haemodynamic instability defined as systolic blood pressure < 90 mmhg or requirement for noradrenaline or adrenaline exceeding 20mcg/minute
* Use of hepatic enzyme inducers, except for phenytoin
* Minor head injury: either normal CT head or not expected to be in intensive care for 72 hours
* GCS = 3 with fixed dilated pupils
* Moribund patient expected to die within 24 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-10; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Core body temperature: bladder temperature probe | 30 minutes after final dose of study drug has been administered

SECONDARY OUTCOMES:
Blood Pressure (systolic and mean arterial pressure) measured by intra-arterial pressure monitor | 6 hourly during study treatment
Liver function test | daily from first dose of study treatment to the 7th day
serum Paracetamol levels (blood analysis) after a single dose of study drug and after final dose of study drug. | baseline, 30, 45, 90, 240 minutes after single dose. 240 minutes after final dose of study drug
Temperature (bladder and tympanic) | Hourly from first study drug treatment until 4 hours after final study drug treatment
  Time-weighted mean, area under the 3-day temperature curve, daily maximum and minimum temperature
The use of physical cooling interventions | hourly during the period of study intervention
Intracranial pressure | 6 hourly during the period of study intervention
  Mean daily intracranial pressure for day 1, 2 and 3.
Incidence of cerebral hypoperfusion | During study intervention period
  1. Systolic blood pressure < 90 mmhg or Mean arterial pressure < 50 mmhg for > 15 minutes
  2. Cerebral perfusion pressure < 50 mmhg for > 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Saxena, Principal Investigator — South East Sydney Illawarra Area Health Service
Locations (2):
- Australia (2):
  - St George Hospital, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland